CLINICAL TRIAL: NCT00410150
Title: A Prospective, Randomized, Controlled, Single Center Trial of the Use of Heliox in Children Admitted to the Hospital With Status Asthmaticus
Brief Title: Heliox-Powered Albuterol Therapy in the Treatment of Children Admitted With Acute Asthma Exacerbation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped after interim analysis and slow enrollment.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Derek Wheeler, Cincinnati Children's Hospital Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-11-34-74-067
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2010-10-13 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-10

CONDITIONS: Status Asthmaticus
Keywords: Status asthmaticus; Asthma; Helium; Children
MeSH Terms: conditions — Status Asthmaticus; Asthma | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Heliox-powered albuterol) (Experimental): Group 1 (Heliox-Powered Albuterol) patients will receive all albuterol nebulizer treatments, including continuous therapy, powered by 70:30 Heliox.
  Interventions: Drug: Helium-oxygen-driven albuterol nebulizer
- Group 2 (Oxygen-powered albuterol) (Active Comparator): Group 2 (Oxygen-Powered Albuterol) patients will receive all albuterol nebulizer treatments, including continuous therapy, powered by 100% oxygen per usual standard of care.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Helium-oxygen-driven albuterol nebulizer — Subjects will be treated with continuous albuterol nebs with Heliox
  Arms: Group 1 (Heliox-powered albuterol)
Drug: Oxygen — Subjects will be treated with continuous albuterol nebs in oxygen
  Arms: Group 2 (Oxygen-powered albuterol)

SUMMARY:
The purpose of this study is to investigate whether heliox-powered albuterol nebulizer therapy will result in reduced inpatient length of stay in children hospitalized with acute asthma exacerbations.

DETAILED DESCRIPTION:
We hypothesize that heliox-powered albuterol nebulizer therapy will result in reduced inpatient length of stay in children hospitalized with acute asthma exacerbations. Severity of asthma will be characterized using a modified Becker Clinical Asthma Score (CAS) based upon the acuity of physical signs for four clinical characteristics (respiratory rate, wheezing, I/E ratio, and accessory muscle use). Scoring will occur at the time of enrollment and every 4 hours thereafter until the patient meets hospital discharge criteria. All scoring using the CAS will be performed by an independent physician, nurse or respiratory therapist blinded to the subject treatment arm. All children will receive standard cardiopulmonary monitoring and treatment, consisting of supplemental oxygen delivered as needed by either nasal cannula or face mask to maintain oxygen saturation >90%, maintenance intravenous fluids, corticosteroid therapy and nebulized albuterol therapy. After written informed consent, eligible children will be randomized to one of two study groups using a sealed envelope technique:

Group 1 (Heliox-Powered Albuterol) patients will receive all albuterol nebulizer treatments, including continuous therapy, powered by 70:30 Heliox.

Group 2 (Oxygen-Powered Albuterol) patients will receive all albuterol nebulizer treatments, including continuous therapy, powered by 100% oxygen per usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 -18 years;
* Previous history of asthma;
* Hospital admission for acute asthma exacerbation;
* Clinical asthma score greater than or equal to 3

Exclusion Criteria:

* Less than 2 years old or over 18 years old;
* Known allergy or hypersensitivity to ß-agonists;
* Require mechanical ventilation (invasive or non-invasive);
* Require FiO2 >0.4;
* Failure to obtain informed consent;
* Enrollment in another investigational drug or asthma protocol;
* Incipient respiratory failure including but limited to respiratory acidosis(pCO2>60 torr), altered mental status and/or excessive work of breathing.

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek S Wheeler, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Rivera ML, Kim TY, Stewart GM, Minasyan L, Brown L. Albuterol nebulized in heliox in the initial ED treatment of pediatric asthma: a blinded, randomized controlled trial. Am J Emerg Med. 2006 Jan;24(1):38-42. doi: 10.1016/j.ajem.2005.06.007. PMID 16338507
- [Background] Kim IK, Phrampus E, Venkataraman S, Pitetti R, Saville A, Corcoran T, Gracely E, Funt N, Thompson A. Helium/oxygen-driven albuterol nebulization in the treatment of children with moderate to severe asthma exacerbations: a randomized, controlled trial. Pediatrics. 2005 Nov;116(5):1127-33. doi: 10.1542/peds.2004-2136. PMID 16263999
- [Background] Bandi V, Velamuri S, Sirgi C, Wendt J, Wendt R, Guntupalli K. Deposition pattern of heliox-driven bronchodilator aerosol in the airways of stable asthmatics. J Asthma. 2005 Sep;42(7):583-6. doi: 10.1080/02770900500216135. PMID 16169793
- [Background] Lee DL, Hsu CW, Lee H, Chang HW, Huang YC. Beneficial effects of albuterol therapy driven by heliox versus by oxygen in severe asthma exacerbation. Acad Emerg Med. 2005 Sep;12(9):820-7. doi: 10.1197/j.aem.2005.04.020. PMID 16141015
- [Background] Ho AM, Lee A, Karmakar MK, Dion PW, Chung DC, Contardi LH. Heliox vs air-oxygen mixtures for the treatment of patients with acute asthma: a systematic overview. Chest. 2003 Mar;123(3):882-90. doi: 10.1378/chest.123.3.882. PMID 12628892
- [Background] Kress JP, Noth I, Gehlbach BK, Barman N, Pohlman AS, Miller A, Morgan S, Hall JB. The utility of albuterol nebulized with heliox during acute asthma exacerbations. Am J Respir Crit Care Med. 2002 May 1;165(9):1317-21. doi: 10.1164/rccm.9907035. PMID 11991886
- [Background] Haynes JM, Sargent RJ, Sweeney EL. Use of heliox to avoid intubation in a child with acute severe asthma and hypercapnia. Am J Crit Care. 2003 Jan;12(1):28-30. No abstract available. PMID 12526234
- [Background] Rose JS, Panacek EA, Miller P. Prospective randomized trial of heliox-driven continuous nebulizers in the treatment of asthma in the emergency department. J Emerg Med. 2002 Feb;22(2):133-7. doi: 10.1016/s0736-4679(01)00454-1. PMID 11858916
- [Background] Dorfman TA, Shipley ER, Burton JH, Jones P, Mette SA. Inhaled heliox does not benefit ED patients with moderate to severe asthma. Am J Emerg Med. 2000 Jul;18(4):495-7. doi: 10.1053/ajem.2000.7365. No abstract available. PMID 10919545
- [Background] Schaeffer EM, Pohlman A, Morgan S, Hall JB. Oxygenation in status asthmaticus improves during ventilation with helium-oxygen. Crit Care Med. 1999 Dec;27(12):2666-70. doi: 10.1097/00003246-199912000-00010. PMID 10628607
- [Background] Kass JE, Terregino CA. The effect of heliox in acute severe asthma: a randomized controlled trial. Chest. 1999 Aug;116(2):296-300. doi: 10.1378/chest.116.2.296. PMID 10453854
- [Background] Henderson SO, Acharya P, Kilaghbian T, Perez J, Korn CS, Chan LS. Use of heliox-driven nebulizer therapy in the treatment of acute asthma. Ann Emerg Med. 1999 Feb;33(2):141-6. doi: 10.1016/s0196-0644(99)70386-0. PMID 9922408
- [Background] Kudukis TM, Manthous CA, Schmidt GA, Hall JB, Wylam ME. Inhaled helium-oxygen revisited: effect of inhaled helium-oxygen during the treatment of status asthmaticus in children. J Pediatr. 1997 Feb;130(2):217-24. doi: 10.1016/s0022-3476(97)70346-9. PMID 9042123
- See also: Cincinnati Children's Hospital Medical Center — http://www.cincinnatichildrens.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Heliox Group: Patients randomized to the Heliox arm of the study
- Control Group: Subjects randomized to the control arm of the study
Period: Overall Study
Arm/Group | Heliox Group | Control Group
Started | 22 | 20
Completed | 20 (2 study withdrawals (analyzed by intention-to-treat)) | 17 (3 study withdrawals (analyzed by intention-to-treat0)
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heliox Group | Control Group | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 20 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.3 (0.8) | 8.2 (0.9) | 7.8 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: Time to discharge eligibility (hours)
Time Frame: Hospital discharge
Measure: Mean (Standard Error); unit: hours
Arm/Group | Heliox Group | Control Group
Number analyzed (Participants) | 22 | 20
hours | 66.2 (8.7) | 63.4 (8.6)

ADVERSE EVENTS:
Arm/Group | Heliox Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No